CLINICAL TRIAL: NCT02217644
Title: Safety, Tolerability and Pharmacokinetics of BI 653048 H3PO4 Oral Drinking Solution in Healthy Male Volunteers (Dose Range: 0.1 mg - 1500 mg). A Singleblind (Within Dose Groups), Randomised, Placebo-controlled Within Dose Groups, Single Rising Dose Phase I Study
Brief Title: Safety, Tolerability and Pharmacokinetics of BI 653048 H3PO4 Oral Drinking Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1262.1
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (4):
- BI 653048 H3PO4 solution (Experimental): single rising doses
  Interventions: Drug: BI 653048 H3PO4 solution
- BI 653048 H3PO4 low dose capsule (Experimental)
  Interventions: Drug: BI 653048 H3PO4 low dose capsule
- BI 653048 H3PO4 high dose capsule (Experimental)
  Interventions: Drug: BI 653048 H3PO4 high dose capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 653048 H3PO4 solution
  Arms: BI 653048 H3PO4 solution
Drug: BI 653048 H3PO4 low dose capsule
  Arms: BI 653048 H3PO4 low dose capsule
Drug: BI 653048 H3PO4 high dose capsule
  Arms: BI 653048 H3PO4 high dose capsule
Drug: Placebo
  Arms: Placebo

SUMMARY:
* Investigation of safety and tolerability of BI 653048 H3PO4 following the administration of single rising doses of an aqueous solution in healthy male subjects
* Pharmacokinetic and pharmacodynamic characteristics of BI 653048, including the investigation of dose proportionality
* Investigation of relative bioavailability of capsules versus aqueous solution

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age ≥21 years and ≤50 years
* Body Mass Index (BMI) ≥18.5 kg/m2 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the trial in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 h) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within 1 week prior to administration or during the trial)
* Any laboratory value outside the reference range that was of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsades des Pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)
* Not willing to use adequate contraception (condom use plus another form of contraception e.g., spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole trial period from the time of the first intake of trial drug until 3 months after the last intake

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant findings in vital signs | up to 10 days after drug administration
  blood pressure (BP), pulse rate (PR) respiratory rate (RR), oral body temperature (T), orthostatic test
Number of patients with clinically significant findings in ECG | up to 10 days after drug administration
Number of patients with clinically significant findings in laboratory tests | up to 10 days after drug administration
Number of patients with adverse events | up to 10 days after drug administration
Assessment of tolerability performed by the investigator on a four-point scale | up to 10 days after drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours after drug administration
tmax (time from dosing to maximum measured concentration) | up to 72 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 72 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after drug administration
AUCt1-t2 (Area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) | up to 72 hours after drug administration
λz (terminal rate constant in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours after drug administration
MRTp.o. (mean residence time of the analyte in the body after oral administration) | up to 72 hours after drug administration
CL/F (total/apparent clearance of the analyte in plasma after extravascular administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 48 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 48 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 48 hours after drug administration
Dose-normalised Cmax | up to 72 hours after drug administration
Dose-normalized AUC0-∞ | up to 72 hours after drug administration
Emax (maximum measured concentration of the biomarker in blood or serum) | up to 72 hours after drug administration
Emin (minimum measured concentration of the biomarker in blood or serum) | up to 72 hours after drug administration
Tmin (time from dosing to minimum measured concentration of the biomarker) | up to 72 hours after drug administration
Tmax (time from dosing to maximum measured concentration of the biomarker) | up to 72 hours after drug administration
AUECt1-t2 (area under the concentration-time curve of the biomarker in the blood over the time interval from t1 to t2) | up to 72 hours after drug administration
AUECbelow_base (area under the baseline corrected concentration-time curve of the biomarker) | up to 72 hours after drug administration
AUECabove_base (area above the baseline corrected concentration-time curve of the biomarker) | up to 72 hours after drug administration
Expression of glucocorticoid responsive genes | up to 72 hours after drug administration

REFERENCES:
- [Derived] Harcken C, Scholl P, Nabozny G, Thomson D, Bianchi D. Clinical profile of the functionally selective glucocorticoid receptor agonist BI 653048 in healthy male subjects. Expert Opin Investig Drugs. 2019 May;28(5):489-496. doi: 10.1080/13543784.2019.1599859. Epub 2019 Apr 9. PMID 30908082